CLINICAL TRIAL: NCT04971785
Title: A Phase 2, Randomized, Double-Blind, Double-Dummy, Placebo-Controlled Study Evaluating the Safety and Efficacy of Semaglutide, and the Fixed-Dose Combination of Cilofexor and Firsocostat, Alone and in Combination, in Subjects With Compensated Cirrhosis (F4) Due to Nonalcoholic Steatohepatitis (NASH)
Brief Title: Study of Semaglutide, and Cilofexor/Firsocostat, Alone and in Combination, in Adults With Cirrhosis Due to Nonalcoholic Steatohepatitis (NASH)
Acronym: WAYFIND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-454-6075; 2021-001445-12 (EudraCT Number); jRCT2071210112 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2021-07-20; First posted 2021-07-21 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — semaglutide; cilofexor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SEMA + CILO/FIR FDC (Experimental): Participants will receive semaglutide (SEMA) 3.0 mg/mL, once weekly and cilofexor and firsocostat (CILO/FIR) 30 mg/20 mg fixed-dose combination (FDC) tablet, once daily up to 72 weeks.
  Interventions: Drug: Semaglutide (SEMA); Drug: Cilofexor (CILO)/Firsocostat (FIR)
- SEMA + PTM CILO/FIR (Experimental): Participants will receive SEMA 3.0 mg/mL, once weekly and Placebo-To-Match (PTM) CILO/FIR FDC tablet, once daily up to 72 weeks.
  Interventions: Drug: Semaglutide (SEMA); Drug: PTM CILO/FIR
- PTM SEMA + CILO/FIR FDC (Experimental): Participants will receive PTM SEMA, once weekly and CILO/FIR 30 mg/20 mg FDC tablet, once daily up to 72 weeks.
  Interventions: Drug: Cilofexor (CILO)/Firsocostat (FIR); Drug: PTM SEMA
- PTM SEMA + PTM CILO/FIR (Placebo Comparator): Participants will receive PTM SEMA, once weekly and PTM CILO/FIR FDC tablet, once daily up to 72 weeks.
  Interventions: Drug: PTM SEMA; Drug: PTM CILO/FIR

INTERVENTIONS:
Drug: Semaglutide (SEMA) — Administered as subcutaneous (SC) injection
  Arms: SEMA + CILO/FIR FDC; SEMA + PTM CILO/FIR
Drug: Cilofexor (CILO)/Firsocostat (FIR) — Tablets administered orally
  Other Names: GS-9674/GS-0976
  Arms: PTM SEMA + CILO/FIR FDC; SEMA + CILO/FIR FDC
Drug: PTM SEMA — Administered as SC injection
  Arms: PTM SEMA + CILO/FIR FDC; PTM SEMA + PTM CILO/FIR
Drug: PTM CILO/FIR — Tablets administered orally
  Arms: PTM SEMA + PTM CILO/FIR; SEMA + PTM CILO/FIR

SUMMARY:
The goal of this clinical study is to understand whether the study drugs, semaglutide (SEMA) with the fixed-dose combination (FDC) of cilofexor/firsocostat (CILO/FIR), cause fibrosis improvement and Nonalcoholic Steatohepatitis (NASH) resolution in participants with cirrhosis due to NASH.

ELIGIBILITY:
Key Inclusion Criteria:

* Liver biopsy consistent with cirrhosis (F4) due to nonalcoholic steatohepatitis (NASH) in the opinion of the central reader. In individuals who have never had a liver biopsy, a screening liver biopsy may be performed.
* Screening laboratory parameters as determined by the study central laboratory:

  * Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m^2, as calculated by the Modification of Diet in Renal Disease (MDRD) equation.
  * Hemoglobin A1c (HbA1c) ≤ 10%
  * International normalized ratio (INR) ≤ 1.4, unless due to therapeutic anticoagulation
  * Platelet count ≥ 125,000/µL
  * Alanine aminotransferase (ALT) < 5 x upper limit of normal (ULN)
  * Serum albumin ≥ 3.5 g/dL
  * Serum alkaline phosphatase (ALP) ≤ 2 x ULN
* Body mass index (BMI) ≥ 23 kg/m^2 at screening.

Key Exclusion Criteria:

* Prior history of decompensated liver disease, including ascites, hepatic encephalopathy (HE), or variceal bleeding.
* Child-Pugh (CP) score > 6 at screening, unless due to an alternative etiology such as Gilbert's syndrome or therapeutic anticoagulation.
* Model for End-stage Liver Disease (MELD) score > 12 at screening, unless due to an alternative etiology such as therapeutic anticoagulation.
* Other causes of liver disease based on medical history and/or central reader review of liver histology, including but not limited to: alcoholic liver disease, autoimmune disorders (eg, primary biliary cholangitis, primary sclerosing cholangitis, autoimmune hepatitis), drug-induced hepatotoxicity, Wilson disease, clinically significant iron overload, or alpha-1-antitrypsin deficiency.
* Chronic hepatitis B virus (HBV) infection (HBsAg positive), or Chronic hepatitis C virus (HCV) infection (HCV antibody and HCV ribonucleic acid (RNA) positive). Individuals cured of HCV infection less than 2 years prior to the screening visit are not eligible.
* History of liver transplantation.
* Current or prior history of hepatocellular carcinoma (HCC).
* Men who habitually drink greater than 21 units/week of alcohol or women who habitually drink greater than 14 units/week of alcohol (1 unit is equivalent to 12 ounce (oz)/360 mL of beer, a 4 oz/120 mL glass of wine, or 1 oz/30 mL of hard liquor).

  * For individuals on vitamin E regimen ≥ 800 IU/day, or pioglitazone, dose must be stable, in the opinion of the investigator for at least 180 days prior to the historical or screening liver biopsy.
  * For individuals on medications for diabetes, dose must be stable, in the opinion of the investigator, for at least 90 days prior to the historical or screening liver biopsy.
* History of type 1 diabetes.
* Treatment with a glucagon-like peptide-1 receptor agonist (GLP-1 RA) in the period from 90 days prior to the screening visit and for individuals with a qualifying historical liver biopsy, for 90 days prior to the date of the historical liver biopsy.
* For individuals who have not completed a series of an authorized coronavirus disease 2019 (COVID-19) vaccination regimen prior to screening, a positive result for COVID-19 on severe acute respiratory syndrome (SARS)-coronavirus 2 (CoV-2) reverse transcriptase-polymerase chain reaction (RT-PCR) test.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (241):
- United States (174):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Digestive Health Specialists, Dothan, Alabama
  - North Alabama Health Research, LLC, Madison, Alabama
  - The Institution For Liver Health dba Arizona Liver Health, Chandler, Arizona
  - Arizona Health Research, Chandler, Arizona
  - The Institute for Liver Health DBA Arizona Liver Health, Peoria, Arizona
  - Gastrointestinal Alliance - Sun City, Sun City, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - The Institution For Liver Health dba Arizona Liver Health, Tucson, Arizona
  - Arkansas Diagnostic Center, Little Rock, Arkansas
  - ARCare Center for Clinical Research, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Southern California Research Center, Coronado, California
  - University of California, San Francisco - Fresno, Fresno, California
  - University of California, San Diego - Altman Clinical and Translational Research Institute, La Jolla, California
  - Gastro Care Institute (Fibroscan), Lancaster, California
  - Digestive Health Research of Southern California, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Keck Medical Center of USC Healthcare Consultation II, Los Angeles, California
  - Biopharma Informatic, LLC, Los Angeles, California
  - United Medical Doctors, Murrieta, California
  - Knowledge Research Center, Orange, California
  - Palmtree Clinical Research, Inc., Palm Springs, California
  - California Liver Research Institute, Pasadena, California
  - Cadena Care Institute, LLC, Poway, California
  - Stanford Medicine Outpatient Center, Redwood City, California
  - Inland Empire Clinical Trials, Rialto, California
  - University of California, Davis Medical Center, Sacramento, California
  - Research and Education Inc., San Diego, California
  - TriWest Research Associates, LLC, San Diego, California
  - Precision Research Institute, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University of California, San Francisco - Liver Clinic, San Francisco, California
  - San Jose Gastroenterology at One Health, San Jose, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - Yale Center for Clinical Investigation, Church Street Research Unit, New Haven, Connecticut
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Synergy Healthcare, Bradenton, Florida
  - Southwest General Healthcare Center, Fort Myers, Florida
  - University of Florida Hepatology Research at the Clinical and Translational Research Building, Gainesville, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Indago Research and Health Center, Inc., Hialeah, Florida
  - Maya Research Center, Hialeah, Florida
  - New Generation of Medical Research, Hialeah, Florida
  - Evolution Clinical Research, INC, Hialeah Gardens, Florida
  - Sunbright Health Medical Center, Homestead, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - UF Health Jacksonville-Gastroenterology Emerson, Jacksonville, Florida
  - Encore Borland-Groover Clinical Research, Jacksonville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - G+C Research Group, Miami, Florida
  - Schiff Center for Liver Diseases/ University of Miami, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Century Research, LLC, Miami, Florida
  - ProLive Medical Research, Corp, Miami, Florida
  - International Medical Investigational Centers, Inc., Miami, Florida
  - Ocean Blue Medical Research Center, Inc, Miami Springs, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Ocala GI Research, Ocala, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Covenant Metabolic Specialists, LLC, Sarasota, Florida
  - Charter Research, Winter Park, Florida
  - Florida Medical Clinic, LLC, Zephyrhills, Florida
  - Southeast Clinical Research LLC, Dalton, Georgia
  - Gastrointestinal (GI) Specialists of Georgia, Marietta, Georgia
  - Rush University Medical Group - Department of Hepatology, Chicago, Illinois
  - Indiana University Health Enterprise Clinical Research Operations, Indianapolis, Indiana
  - Gastroenterology Health Partners, PLLC, New Albany, Indiana
  - Digestive Research Alliance of Michigan, South Bend, Indiana
  - Iowa Digestive Disease Center, PC, Clive, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kansas Medical Clinic PA, Topeka, Kansas
  - GI Alliance, Baton Rouge, Louisiana
  - Combined Gastro Research, LLC, Lafayette, Louisiana
  - Tandem Clinical Research GI, LLC, Marrero, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Oschner Clinic Foundation, New Orleans, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Woodholme Gastroenterology Associates, Glen Burnie, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Greater Boston Gastroenterology, Framingham, Massachusetts
  - Hawthorn Medical Associates, South Dartmouth, Massachusetts
  - Michigan Medicine - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinical Research Center, Wyoming, Michigan
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - GI Alliance, Flowood, Mississippi
  - Southern Therapy and Advanced Research, Jackson, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - GI Associates Research, Columbia, Missouri
  - Kansas City Research Institute, Kansas City, Missouri
  - Sierra Clinical Research, Las Vegas, Nevada
  - Digestive Disease Research, Florham Park, New Jersey
  - Allied Health Clinical Research Organization, LLC, Freehold, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Center for Research at Southwest Gastroenterology Associates, PC, Albuquerque, New Mexico
  - Northwell Health Center for Liver Diseases, Manhasset, New York
  - New York University Langone Health, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Liver Clinic (study visits, Fibroscan): Columbia University Irving Medical Center / NewYork Presbyterian Hospital, New York, New York
  - The New York - Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Asheville Gastroenterology, a Division of Digestive Health Partners, PA, Asheville, North Carolina
  - Atrium Health Transplant and Center for Liver Disease, Charlotte, North Carolina
  - Charlotte Gastroenterology & Hepatology, PLLC, Charlotte, North Carolina
  - Northeast GI Research Division, Concord, North Carolina
  - Coastal Research Institute, Fayetteville, North Carolina
  - Lucas Research, Inc., Morehead City, North Carolina
  - Carolina's GI Research, LLC, Raleigh, North Carolina
  - Optimed Research, Columbus, Ohio
  - DSI Research, Springboro, Ohio
  - Clinical Research Institute of Ohio, LLC, Westlake, Ohio
  - Options Health Research, LLC, Tulsa, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - University Gastroenterology, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Columbia Digestive Health Research, Columbia, South Carolina
  - Digestive Disease Research Center, Greenwood, South Carolina
  - Velocity Clinical Research, Spartanburg, Spartanburg, South Carolina
  - Wake Research - ClinsSearch, LLC, Chattanooga, Tennessee
  - Gastrointestinal Associates of Northeast Tennessee, Johnson City, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Pinnacle Clinical Research, Austin, Texas
  - South Texas Research Institute, Brownsville, Texas
  - GI Alliance, Cedar Park, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - GI Alliance, Dallas, Texas
  - Internal Medicine Digestive and Liver Diseases Clinical Trials, Dallas, Texas
  - Soma Clinical Trials, LLC, Denison, Texas
  - DHR Health Institute for Research and Development Cancer Research Center, Edinburg, Texas
  - South Texas Research Institute, Edinburg, Texas
  - GI Alliance, Fort Worth, Texas
  - GI Alliance, Garland, Texas
  - Pinnacle Clinical Research, Georgetown, Texas
  - Texas Digestive Specialists, Harlingen, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Liver Associates of Texas, P.A., Houston, Texas
  - Liver Specialists of Texas, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Houston Research Institute, Houston, Texas
  - BioStar Clinical Research Group Inc., Katy, Texas
  - GI Alliance, Lubbock, Texas
  - Biopharma Informatic, LLC, McAllen, Texas
  - Digestive System Healthcare, Pasadena, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Diabetes and Glandular Disease Clinic, P.A., San Antonio, Texas
  - Pinnacle Clinical Research, LLC, San Antonio, Texas
  - GI Alliance (Patients Seen, IP Shipment & Fibroscan), San Marcos, Texas
  - Impact Research Institute, Waco, Texas
  - GI Alliance, Webster, Texas
  - Digestive Health Research of North Texas, Wichita Falls, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - The University Of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours Richmond Community Hospital, Inc. d/b/a Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - Virginia Commonwealth University Health Clinical Research Services Unit, Richmond, Virginia
  - Virginia Mason, Seattle, Washington
  - Liver Institute Northwest, Seattle, Washington
- Australia (7):
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Eastern Health, Box Hill Hospital, Box Hill, Victoria
  - Monash Health, Monash Medical Centre (Clayton), Clayton, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Canada (11):
  - Wlliam Osler Health System - Brampton Civic Hospital, Brampton
  - University of Calgary Liver Unit - Heritage Medical Research Clinic, Calgary
  - McMaster University Medical Center, Hamilton
  - London Health Sciences Centre - University Hospital, London
  - Centre de Recherche du Centre Hospitalier de I'Universite de Montreal (CRCHUM), Montreal
  - Chronic Viral Illness Service, Royal Victoria Hospital, McGill University Health Centre (MUHC), Montreal
  - Toronto General Hospital - University Health Network, Toronto
  - Toronto Liver Centre, Toronto
  - Gordon and Leslie Diamond Health Care Centre, Vancouver General Hospital, UBC Division of Gastroenterology, Vancouver
  - (G.I.R.I.) Gastrointestinal Research Institute, Vancouver
  - Toronto Digestive Disease Associates Specialty Research, Vanghan
- France (18):
  - CHU Amiens Picardie, Amiens
  - Centre Hosptitalier Universitaire d'Angers, Angers
  - Centre Hospitalier Regional Universitaire de Tours - Hopital Trousseau, Chambray-lès-Tours
  - Hopital Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Hopital Claude Huriez, Lille
  - Centre Hospitalier Universitaire Limoges, Limoges
  - Hopital de la Croix-Rousse, Lyon
  - Hopital Saint Joseph, Marseille
  - Centre Hospitalier Universitarie de Montpellier - Hospital Saint-Eloi, Montpellier
  - Centre Hospitalier Universitaire de Nice - Hopital L'archet, Nice
  - Hopital Universitaire Pitie Salpetriere, Paris
  - Hopitaux de Paris - Hopital Cochin, Paris
  - Hopital Beaujon, Pessac
  - Hopital Haut Leveque, Pessac
  - CHU Rennes Pontchaillou, Rennes
  - Hopital Rangueil, Toulouse
  - Hopital Brabois Adultes - CHU de Nancy, Vandœuvre-lès-Nancy
- Japan (12):
  - Fukui-ken Saiseikai Hospital, Fukui
  - Juntendo University Shizouka Hospital, Izunokuni
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Japanese Red Cross Masashino Hospital, Musashino
  - Osaka City University Hospital, Osaka
  - Saga University Hospital, Saga
  - Sapporo-Kosei General Hospital, Sapporo
  - Saiseikai Suita Hospital, Suita
  - Federation of National Public Service Personnel Mutual Aid Associations Toranomon Hospital, Tokyo
  - Ehime University Hospital, Toon-Shi
  - Yamagata University Hospital, Yamagata
  - Yokohama City University Hospital, Yokohama
- Puerto Rico (3):
  - Latin Clinical Trial Center, San Juan
  - VA Caribbean Healthcare System, San Juan
  - FDI Clinical Research, San Juan
- Spain (16):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Torrecardenas, Almería
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic De Barcelona, Barcelona
  - Hospital General Universiatrio Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz Edificio de Malemidad, Madrid
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgin del Rocio, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario y Politecnlo la Fe, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-454-6075

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Canada, France, Japan, Australia and Spain.
Pre-assignment Details: 1595 participants were screened.
Groups:
- SEMA + CILO/FIR FDC: Participants received semaglutide (SEMA) 3.0 mg/mL subcutaneous (SC) injection once weekly and cilofexor and firsocostat (CILO/FIR) 30 mg/20 mg fixed-dose combination (FDC) tablet orally, once daily up to 72 weeks.
- SEMA + PTM CILO/FIR: Participants received SEMA 3.0 mg/mL SC injection, once weekly and Placebo-To-Match (PTM) CILO/FIR FDC tablet orally, once daily up to 72 weeks.
- PTM SEMA + CILO/FIR FDC: Participants received PTM SEMA SC injection, once weekly and CILO/FIR 30 mg/20 mg FDC tablet orally, once daily up to 72 weeks.
- PTM SEMA + PTM CILO/FIR: Participants received PTM SEMA SC injection, once weekly and PTM CILO/FIR FDC tablet orally, once daily up to 72 weeks.
Period: Overall Study
Arm/Group | SEMA + CILO/FIR FDC | SEMA + PTM CILO/FIR | PTM SEMA + CILO/FIR FDC | PTM SEMA + PTM CILO/FIR
Started | 125 | 124 | 123 | 85
Completed | 103 | 104 | 91 | 65
Not Completed | 22 | 20 | 32 | 20
Not completed — Withdrew Consent | 5 | 5 | 17 | 7
Not completed — Adverse Event | 7 | 8 | 6 | 3
Not completed — Lost to Follow-up | 2 | 1 | 6 | 7
Not completed — Protocol Violation | 3 | 1 | 1 | 2
Not completed — Investigator's Discretion | 3 | 1 | 1 | 0
Not completed — Randomized but Never Treated | 1 | 2 | 0 | 1
Not completed — Death | 0 | 1 | 1 | 0
Not completed — Site Terminated by Sponsor | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | SEMA + CILO/FIR FDC | SEMA + PTM CILO/FIR | PTM SEMA + CILO/FIR FDC | PTM SEMA + PTM CILO/FIR | Total
Number analyzed (Participants) | 124 | 122 | 123 | 84 | 453
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 72 | 73 | 67 | 44 | 256
  >=65 years | 52 | 49 | 56 | 40 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (10.4) | 61 (9.2) | 62 (9.5) | 63 (9.1) | 62 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 85 | 74 | 50 | 292
  Male | 41 | 37 | 49 | 34 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 23 | 30 | 19 | 100
  Not Hispanic or Latino | 95 | 99 | 90 | 62 | 346
  Unknown or Not Reported | 1 | 0 | 3 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 1 | 2 | 7
  Asian | 11 | 9 | 15 | 3 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 5 | 9
  White | 100 | 108 | 98 | 66 | 372
  More than one race | 5 | 2 | 3 | 4 | 14
  Unknown or Not Reported | 3 | 1 | 5 | 4 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 95 | 99 | 88 | 63 | 345
  Canada | 7 | 7 | 12 | 6 | 32
  France | 5 | 5 | 9 | 10 | 29
  Japan | 4 | 6 | 6 | 1 | 17
  Australia | 6 | 2 | 6 | 2 | 16
  Spain | 7 | 3 | 2 | 2 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved ≥ 1-Stage Improvement in Fibrosis Without Worsening of Nonalcoholic Steatohepatitis (NASH) at Week 72 in Semaglutide (SEMA) + Cilofexor/Firsocostat (CILO/FIR) Fixed Dose Combination (FDC) Versus Placebo Groups
Description: Fibrosis improvement was defined as ≥ 1-stage decrease from baseline in fibrosis according to the NASH clinical research network (CRN) classification. Worsening of NASH was defined as ≥ 1-point increase from baseline in hepatocellular ballooning or lobular inflammation.
  Clopper-Pearson method was used in outcome measure analysis in each arm. Percentages were rounded-off.
Time Frame: Week 72
Population: Participants in the Full Analysis Set in SEMA + CILO/FIR FDC and PTM SEMA + PTM CILO/FIR were analyzed. The Full Analysis Set included all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SEMA + CILO/FIR FDC | PTM SEMA + PTM CILO/FIR
Number analyzed (Participants) | 124 | 84
percentage of participants | 13.7 [8.2 to 21.0] | 8.3 [3.4 to 16.4]
Statistical Analysis 1: Comparison: SEMA + CILO/FIR FDC vs PTM SEMA + PTM CILO/FIR; Test type: Superiority; p = 0.2289, Stratified Mantel-Haenszel test; Difference in percentages = 5.7, 95% CI 2-sided [-3.6 to 14.9] — Percentage difference and 95% confidence interval (CI) between each pair of treatment groups were from stratified Mantel-Haenszel test with baseline diabetes status and baseline enhanced liver fibrosis (ELF) category as stratification factors

2. Secondary Outcome: Percentage of Participants Who Achieved ≥1-Stage Improvement in Fibrosis Without Worsening of NASH at Week 72 in SEMA + CILO/FIR FDC Versus SEMA Alone
Description: Fibrosis improvement was defined as ≥ 1-stage decrease from baseline in fibrosis according to the NASH CRN classification. Worsening of NASH was defined as ≥ 1-point increase from baseline in hepatocellular ballooning or lobular inflammation.
  Clopper-Pearson method was used in outcome measure analysis in each arm. Percentages were rounded-off.
Time Frame: Week 72
Population: Participants in the Full Analysis Set in SEMA + CILO/FIR and SEMA + PTM CILO/FIR were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SEMA + CILO/FIR FDC | SEMA + PTM CILO/FIR
Number analyzed (Participants) | 124 | 122
percentage of participants | 13.7 [8.2 to 21.0] | 15.6 [9.6 to 23.2]
Statistical Analysis 1: Comparison: SEMA + CILO/FIR FDC vs SEMA + PTM CILO/FIR; Test type: Superiority; p = 0.6959, Stratified Mantel-Haenszel test; Difference in percentages = -1.8, 95% CI 2-sided [-11.1 to 7.4] — Percentage difference and 95% CI between each pair of treatment groups presented were from stratified Mantel-Haenszel test with baseline diabetes status and baseline ELF category as stratification factors

3. Secondary Outcome: Percentage of Participants With NASH Resolution Without Worsening in Fibrosis at Week 72 in SEMA + CILO/FIR FDC Versus Placebo Groups
Description: NASH resolution is defined as lobular inflammation of 0 or 1 and hepatocellular ballooning of 0. Worsening in fibrosis was defined as a change in fibrosis worsening stage as per NASH CRN criteria.
  Clopper-Pearson method was used in outcome measure analysis in each arm. Percentages were rounded-off.
Time Frame: Week 72
Population: Participants in the Full Analysis Set in SEMA + CILO/FIR FDC and PTM SEMA + PTM CILO/FIR with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SEMA + CILO/FIR FDC | PTM SEMA + PTM CILO/FIR
Number analyzed (Participants) | 82 | 49
percentage of participants | 57.3 [45.9 to 68.2] | 22.4 [11.8 to 36.6]
Statistical Analysis 1: Comparison: SEMA + CILO/FIR FDC vs PTM SEMA + PTM CILO/FIR; Test type: Superiority; p < 0.0001, Stratified Mantel-Haenszel test; Difference in percentages = 35.7, 95% CI 2-sided [18.8 to 52.6] — Percentage difference and 95% CI between each pair of treatment groups presented are from stratified Mantel-Haenszel test with baseline diabetes status and baseline ELF category as stratification factors

4. Secondary Outcome: Percentage of Participants With NASH Resolution Without Worsening in Fibrosis In Participants Treated With SEMA + CILO/FIR FDC Versus CILO/FIR Alone Groups
Description: as for outcome 3
Time Frame: Week 72
Population: Participants in the Full Analysis Set in SEMA + CILO/FIR FDC and PTM SEMA + CILO/FIR FDC with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SEMA + CILO/FIR FDC | PTM SEMA + CILO/FIR FDC
Number analyzed (Participants) | 82 | 88
percentage of participants | 57.3 [45.9 to 68.2] | 31.8 [22.3 to 42.6]
Statistical Analysis 1: Comparison: SEMA + CILO/FIR FDC vs PTM SEMA + CILO/FIR FDC; Test type: Superiority; p = 0.0006, Stratified Mantel-Haenszel test; Difference in percentages = 26.1, 95% CI 2-sided [11.3 to 40.9] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: All-cause mortality and Adverse events: Up to 72 weeks plus 35 days
Description: All-cause mortality: The All Randomized Analysis Set included all participants who were randomized in the study.
  Adverse events: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | SEMA + CILO/FIR FDC | SEMA + PTM CILO/FIR | PTM SEMA + CILO/FIR FDC | PTM SEMA + PTM CILO/FIR
All-Cause Mortality (participants affected / at risk) | 0/125 | 1/124 | 1/123 | 0/85
Serious Adverse Events (participants affected / at risk) | 17/124 | 13/122 | 18/123 | 11/84
Other Adverse Events (participants affected / at risk) | 101/124 | 97/122 | 85/123 | 60/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SEMA + CILO/FIR FDC (N=124) | SEMA + PTM CILO/FIR (N=122) | PTM SEMA + CILO/FIR FDC (N=123) | PTM SEMA + PTM CILO/FIR (N=84)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Prosthetic cardiac valve stenosis (General disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 1 | 0
Covid-19 pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 0 | 0 | 0 | 1
Large intestine infection (Infections and infestations) | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Shoulder fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Diffuse idiopathic skeletal hyperostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 3 | 1
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Sensory loss (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 3 | 0 | 0 | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SEMA + CILO/FIR FDC (N=124) | SEMA + PTM CILO/FIR (N=122) | PTM SEMA + CILO/FIR FDC (N=123) | PTM SEMA + PTM CILO/FIR (N=84)
Abdominal distension (Gastrointestinal disorders) | 9 | 10 | 4 | 6
Abdominal pain (Gastrointestinal disorders) | 11 | 10 | 6 | 11
Abdominal pain upper (Gastrointestinal disorders) | 7 | 11 | 6 | 8
Constipation (Gastrointestinal disorders) | 30 | 26 | 11 | 7
Diarrhoea (Gastrointestinal disorders) | 34 | 25 | 16 | 15
Dyspepsia (Gastrointestinal disorders) | 12 | 2 | 4 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 13 | 3 | 2
Nausea (Gastrointestinal disorders) | 59 | 49 | 29 | 19
Vomiting (Gastrointestinal disorders) | 27 | 21 | 7 | 6
Fatigue (General disorders) | 17 | 17 | 9 | 11
Bronchitis (Infections and infestations) | 2 | 3 | 5 | 5
Covid-19 (Infections and infestations) | 21 | 15 | 15 | 14
Influenza (Infections and infestations) | 1 | 2 | 3 | 5
Nasopharyngitis (Infections and infestations) | 7 | 4 | 6 | 4
Sinusitis (Infections and infestations) | 8 | 8 | 4 | 6
Upper respiratory tract infection (Infections and infestations) | 7 | 4 | 12 | 4
Urinary tract infection (Infections and infestations) | 13 | 6 | 8 | 3
Decreased appetite (Metabolism and nutrition disorders) | 19 | 20 | 7 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 7 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 14 | 4 | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 6 | 12 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7 | 8 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 7 | 3
Dizziness (Nervous system disorders) | 7 | 10 | 9 | 8
Headache (Nervous system disorders) | 7 | 11 | 12 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 7 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 13 | 12 | 6
Hypertension (Vascular disorders) | 3 | 1 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years.

DOCUMENTS (2):
  • Study Protocol (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT04971785/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT04971785/SAP_001.pdf